CLINICAL TRIAL: NCT06388824
Title: The Effect of a Single Low Dose of Esketamine During Surgical Abortion in Patients With Sleep Disturbance
Brief Title: The Effect of Esketamine on Sleep Disturbance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWang028
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Sleep Disturbance
Keywords: Esketamine; surgical abortion
MeSH Terms: conditions — Parasomnias | interventions — Saline Solution; Sodium Chloride; Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group of patients undergoing surgical abortion with normal saline (Placebo Comparator): Patients undergoing surgical abortion received a single injection of 5ml 0.9% normal saline after the beginning of surgery
  Interventions: Drug: normal saline
- Group of patients undergoing surgical abortion with esketamine (Active Comparator): Patients undergoing surgical abortion received a single injection of 0.2mg/kg esketamine after the beginning of surgery
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: normal saline — Patients undergoing surgical abortion received a single injection of 5ml 0.9% normal saline after the beginning of surgery
  Other Names: sodium chloride injection
  Arms: Placebo Group of patients undergoing surgical abortion with normal saline
Drug: Esketamine — Patients undergoing surgical abortion received a single injection of 0.2mg/kg esketamine after the beginning of surgery
  Other Names: Esketamine Hydrochloride Injection
  Arms: Group of patients undergoing surgical abortion with esketamine

SUMMARY:
To explore the efficacy of a single low dose of esketamine during surgical abortion in patients with sleep disturbance

DETAILED DESCRIPTION:
Sleep disturbance occur in the form of sleep deprivation, circadian rhythm disturbance, and structural abnormalities. Women who requires surgical abortion due to fetal anomaly or unwanted pregnancy often experience sleep disturbance. Severe sleep disturbance is a strong indicator for postoperative sleep disorders, which can lead to postoperative delirium and cognitive dysfunction, aggravate postoperative pain, and delay postoperative recovery.

Esketamine is an N-methyl-D-aspartate(NMDA) receptor antagonist with analgesic and sedative effects, and is widely used in clinical treatment of refractory depression. For patients undergoing surgical abortion, in addition to sedation and analgesia, whether the intraoperative use of esketamine has positive effects on sleep disturbance is worth exploring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older with sleep disturbance;
2. American Society of Anesthesiologists physical status I-III;
3. A gestational age below 12 weeks;
4. Elective surgery is proposed;
5. BMI of 19-30 kg/m2;
6. Patients who agreed to enroll in this study voluntarily

Exclusion Criteria:

1. Any contraindications to ketamine or esketamine;
2. Allergic history of general anesthesia drugs, opioid drugs, non-steroidal drugs;
3. Respiratory insufficiency, respiratory failure;
4. Bronchial asthma, severe hypertension, severe hepatic and renal dysfunction, severe cardiovascular disease, or hyperthyroidism;
5. BMI<18 kg/m2 or BMI>30kg/m2;
6. Poor compliance, unable to complete the experiment according to the study plan; Participants who have participated in clinical trials of other drugs within the last 4 weeks;
7. Any circumstances deemed unsuitable for inclusion by the researcher for any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
The incidence of sleep disturbance on the first night after surgery | the first night after surgery
  Patients completed the sleep quality scale (AIS, Athens Insomnia Scale) on the first night after surgery. The AIS has a total of 8 items,with scores ranging from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.We asked the patients to fill out this questionnaire after the first postoperative night to evaluate the changes in sleep quality. We recorded AIS scores as statistical indicators.

SECONDARY OUTCOMES:
The incidence of sleep disturbance on the second and third postoperative nights | the second and third nights after surgery
  Patients completed the sleep quality scale(AIS, Athens Insomnia Scale) on the second and third day after surgery. The AIS has a total of 8 items,with scores ranging from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.We asked the patients to fill out this questionnaire after the second and third postoperative nights to evaluate the changes in sleep quality. We recorded AIS scores as statistical indicators.
The incidence of sleep disturbance on the seventh postoperative nights | the seventh night after surgery
  Patients completed the sleep quality scale(AIS, Athens Insomnia Scale) on the seventh day after surgery. The AIS has a total of 8 items,with scores ranging from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.We asked the patients to fill out this questionnaire after the seventh postoperative nights to evaluate the changes in sleep quality. We recorded AIS scores as statistical indicators.
Postoperative anxiety | 1 day before surgery, 1, 2, 3 and 7 days after surgery
  Patients completed the anxiety rating scales (HADS-A,Hospital Anxiety and Depression Scale-Anxiety subscale) on the day before surgery. HADS-A consists of 7 items, each question in the questionnaire was scored on a scale of 0-3, and a total score of 8 points or higher is diagnosed as anxiety. And we asked the patients to fill out this questionnaire on the 1, 2, 3 and 7 days after surgery again to evaluate the changes in anxiety. We recorded HADS-A scores as statistical indicators.
Postoperative depression | 1 day before surgery, 1, 2, 3 and 7 days after surgery
  Patients completed the depression rating scales (HADS-D,Hospital Anxiety and Depression Scale-Depression subscale) on the day before surgery. HADS-D consists of 7 items, each question in the questionnaire was scored on a scale of 0-3, and a total score of 8 points or higher is diagnosed as depression. And we asked the patients to fill out this questionnaire on the 1, 2, 3 and 7 days after surgery again to evaluate the changes in depression. We recorded HADS-D scores as statistical indicators.
Pain intensity | 1 hour after surgery, 1, 2, 3 and 7 days after surgery
  The pain score at rest or after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
Adverse event | Within 1 hour after surgery, within 1 day after surgery
  All kinds of adverse events (nausea, vomiting, tachycardia, hypertension, somnolence, dizziness, hallucination, diplopia, etc) occurred in patients were recorded
preoperative hemoglobin concentration | the day before surgery
  Hemoglobin concentration in venous blood was measured.
Human Chorionic Gonadotropin level | within one week before surgery, within one week after surgery
  Human Chorionic Gonadotropin (HCG) in venous blood was measured.
The incidence of sleep disturbance on the day before surgery | the day before surgery
  Patients completed the sleep quality scale (AIS, Athens Insomnia Scale) on the day before surgery. The AIS has a total of 8 items,with scores ranging from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.We asked the patients to fill out this questionnaire on the day before surgery to evaluate the changes in sleep quality. We recorded AIS scores as statistical indicators.
The incidence of sleep disturbance before surgery | the day before surgery
  Patients completed the sleep quality scale (PSQI, Pittsburgh sleep quality index) on the day before surgery. The PSQI has a total of 24 items(Including 19 self-evaluation items and 5 other evaluation items),of which the 19th self-evaluation item and 5 other self-evaluation items do not participate in scoring, while the remaining 18 self-evaluation items participate in scoring, with each item scoring 0-3 points. The total score of the scale ranges from 0 to 21 points, with a total score higher than 5 indicating poor sleep quality. We require patients to fill out this questionnaire one day before surgery to evaluate whether they have had sleep disorders in the past month.We recorded PSQI scores as statistical indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, PhD, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Z, Miao M, Huang F, Hu L, Yang X, Cui W, Yu Y, Wang G, Wang C, Zhang L. Effect of a single low-dose esketamine administration during surgical abortion on postoperative sleep disturbance: a randomized controlled trial. Nat Commun. 2025 Aug 14;16(1):7533. doi: 10.1038/s41467-025-62933-1. PMID 40804260